CLINICAL TRIAL: NCT02842333
Title: Study of Predictive Immunological Parameters of Molecular Complete Remission in Patients With Chronic Myelogenous Leukemia in Chronic Phase and Treated With Tyrosine Kinase Inhibitor
Acronym: PAMIR01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2015/263
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2023-04

CONDITIONS: Chronic Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Additional biological samples (Experimental): Blood samples will be realized at inclusion and 6 months after inclusion (optional).
  Peripheral Blood Mononuclear Cells (PBMC) will be collected.
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — Blood samples

SUMMARY:
The investigators recently identified promiscuous HLA-DR-derived epitopes from the human telomerase reverse transcriptase (TERT) called universal cancer peptides (UCP), to study tumor-specific CD4+ T cell responses.

The aim of this prospective preliminary study is to evaluate the presence of UCP-specific Th1 responses in patients in complete remission of CML two years after end of Tyrosine Kinase Inhibitor (TKi) treatments.

ELIGIBILITY:
Inclusion Criteria:

* For cohort A :

  * patient with chronic myelogenous leukemia in chronic phase in deep molecular response (MR4.0) persistent for 2 years or more after end of TKi treatments
  * patient with total cessation of TKi treatment
  * signed written informed consent
* For cohort B :

  * patient with chronic myelogenous leukemia in chronic phase, for whom a diagnosis of relapse was increased 1 year or less after stopping treatment with TKIs (inclusion of patient under TKi treatment after relapse is possible).
  * signed written informed consent

Exclusion Criteria (for all patients) :

* patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (corticoids ≤ 10 mg/day is allowed)
* active autoimmune diseases, HIV, hepatitis C or B virus
* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study.
* patient under guardianship, curator or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
UCP-specific Th1 responses measured by ELISPOT assay | at inclusion

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - CHU de Dijon, Dijon
  - CHU de Nice, Nice
  - Hôpital Saint-Louis, Paris

IPD SHARING:
Plan to Share IPD: No